CLINICAL TRIAL: NCT00434395
Title: A Randomized, Double-Blind, Placebo- and Moxifloxacin (Open-Label)-Controlled, 4-Period Crossover Study of the Effects of a Single Dose of MOA-728 Infused Intravenously on Cardiac Repolarization in Healthy Subjects
Brief Title: Study Evaluating the Effects of MOA-728 on Cardiac Repolarization in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3200L2-104
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Healthy

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
The purpose of the study is to assess the effects of MOA-728 on cardiac repolarization in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy subjects men or women aged 18-50

Exclusion Criteria:

* Any significant clinically important disease
* Family history of long QT syndrome and/or sudden cardiac death
* Allergy to moxifloxacin or the quinolone class of antibiotics

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-03; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Cardiac repolarization will be assessed by the QTc interval in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Phoenix, Arizona, United States